CLINICAL TRIAL: NCT06718257
Title: Chemotherapy Combined with Immunotherapy and Targeted Therapy in Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Chemotherapy Combined with Immunotherapy and Targeted Therapy in Cholangiocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1058
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Cholangiocarcinoma
Keywords: advanced cholangiocarcinoma; chemotherapy combined with immunotherapy and targeted therapy; clinical efficacy and safety
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Patients initially received GP/GEMOX regimen.
  Interventions: Drug: Gemcitabine combined with cisplatin or oxaliplatin
- Experimental group: Patients initially received GP/GEMOX combined with PD-1/L1 and TKI inhibitors regimen.
  Interventions: Drug: Gemcitabine combined with cisplatin or oxaliplatin, PD-1/L1 and TKI inhibitors

INTERVENTIONS:
Drug: Gemcitabine combined with cisplatin or oxaliplatin — Gemcitabine (1000 mg/m², day 1 and 8) and cisplatin (75 mg/m², day 1) or oxaliplatin (85 mg/m², day 1)
  Groups: Control group
Drug: Gemcitabine combined with cisplatin or oxaliplatin, PD-1/L1 and TKI inhibitors — Gemcitabine (1000 mg/m², day 1 and 8), cisplatin (75 mg/m²; day 1) or oxaliplatin (85 mg/m²; day 1), PD-1/L1 agents (200 mg; day 1), and TKI inhibitors (8 mg; per day)
  Groups: Experimental group

SUMMARY:
This study aims to validate the efficacy and safety of GP/GEMOX combined with PD-1/L1 inhibitors and TKI agents in patients with advanced cholangiocarcinoma through a multicenter, retrospective study to guide clinical practice.

DETAILED DESCRIPTION:
This study plans to enroll patients diagnosed with advanced cholangiocarcinoma. After confirming patients treated with GP/GEMOX or GP/GEMOX combined with PD-1/L1 and TKI agents as initial therapy, the investigators will collect relevant clinical data, including basic clinical information, laboratory data, imaging data, pathological data, and surgical data through an electronic medical record system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiologically confirmed intrahepatic cholangiocarcinoma
* Initially treated with GP/GEMOX or GP/GEMOX combined with PD-1/L1 and TKI inhibitors

Exclusion Criteria:

* Direct surgery after hospitalization
* Initial treatment combined with local therapies (radiotherapy, radiofrequency, particle implantation, TACE, etc.)
* Initial treatment involving other comprehensive therapeutic regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were histologically or radiologically confirmed intrahepatic cholangiocarcinoma, with initial treatment consisting of GP/GEMOX or GP/GEMOX combined with PD-1/L1 and TKI inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 1 year
  Overall survival (OS) is defined as the time from cancer diagnosis to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS) is defined as the time from the start of treatment until disease progression or the emergence of new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, PHD, Study Chair — Department of Hepatobiliary and Pancreatic Surgery, Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided